CLINICAL TRIAL: NCT05938712
Title: A Two Arm, Open Label, Pilot Study to Evaluate the Safety and Efficacy of the Combined Use of Once Daily 10mg Dapagliflozin and Once Weekly 1.0mg Semaglutide in Kidney Transplant Recipients
Brief Title: The Efficacy, Mechanism & Safety of Sodium Glucose Co-Transporter-2 Inhibitor & Glucagon-Like Peptide 1 Receptor Agonist Combination Therapy in Kidney Transplant Recipients
Acronym: HALLMARK
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Sunita Singh, MD, MSc, FRCPC, Clinician Scientist, University Health Network, Toronto
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 23-5050
Record Dates: First submitted 2023-05-16; First posted 2023-07-10 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Kidney Transplant Recipients
Keywords: Type 2 diabetes; SGLT2 inhibition; GLP-1 receptor agonist
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; semaglutide

STUDY DESIGN:
Intervention Model Description: Patients will be allocated to treatment with either dapagliflozin 10 mg PO daily alone for 12 weeks or subcutaneous once weekly semaglutide up-titrated as tolerated every 4 weeks starting with 0.25 mg, then to 0.5 mg to 1 mg alone for 12 weeks, followed by a subsequent treatment period of combination therapy with dapagliflozin 10 mg PO daily plus maximally tolerated dose semaglutide (up-titrated every 4 weeks from 0.25 mg to 0.5 mg to 1 mg) subcutaneous once weekly.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental): Semaglutide Subcutaneous 0.25mg once weekly for 4 weeks, then 0.5mg once weekly for 4 weeks, then 1mg once weekly for 4 weeks.
  Interventions: Drug: Dapagliflozin 10 MG; Drug: Semaglutide, 1.0 mg/mL
- Dapagliflozin (Experimental): Dapagliflozin Tablets Total Dose 10mg daily for 12 weeks
  Interventions: Drug: Dapagliflozin 10 MG; Drug: Semaglutide, 1.0 mg/mL

INTERVENTIONS:
Drug: Dapagliflozin 10 MG — Semaglutide subcutaneous once weekly for 12 weeks.
  Other Names: FARXIGA
Drug: Semaglutide, 1.0 mg/mL — Dapagliflozin oral once daily for 12 weeks.
  Other Names: OZEMPIC

SUMMARY:
The study aims to determine the short-term efficacy, mechanisms and safety of 12 weeks of dapagliflozin and semaglutide combination therapy in 20 KTR, with and without T2D.

DETAILED DESCRIPTION:
Kidney transplantation improves survival and quality of life for patients with kidney failure. However, treatment options to protect the heart and the kidney in transplant recipients are lacking. Sodium-glucose cotransporter 2 (SGLT2) inhibitors and glucagon-like peptide-1 receptor agonists (GLP-1RA) are novel anti-diabetic drugs which not only lower blood sugar, but also lower blood pressure in the kidney's individual filtering units and protect kidney function in the long term. It is unclear if the protective mechanisms of these drugs also occur in people with a kidney transplant. Several smaller studies have shown that SGLT2 inhibitors or GLP-1RA used alone are safe in people with kidney transplants. No studies have yet to look at the combined use of SGLT2 inhibitors and GLP-1RA in kidney transplant recipients (KTR).

The purpose of the HALLMARK study is to determine the mechanisms and safety of the combination use of semaglutide, a GLP-1RA, and dapagliflozin, a SGLT2 inhibitor. To investigate this, 20 kidney transplant recipients with and without diabetes will be treated with both semaglutide or dapagliflozin for 12 weeks followed by a combination of semaglutide and dapagliflozin for 12 weeks. The study will measure salt and water removal as well as the effect on blood pressure, kidney function, heart function, liver stiffness as well as the safety of these agents.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent.
* Patients aged ≥18 years with KTR
* >3 months post kidney transplantation
* Estimated glomerular filtration rate [eGFR] ≥20 ml/min/1.73m2
* BP <160/100 and >90/60 at screening
* Body-mass index [BMI] between 18.5-40kg/m2
* In patients with T2D or PTDM, HbA1c <12.0%;

Exclusion Criteria:

* Type 1 diabetes.
* History of multi-organ transplant
* Acute coronary syndrome, transient ischemic attack or stroke within 30 days prior to screening
* Impending need for kidney biopsy or rapid decline in eGFR within 30 days prior to screening
* Actively treated BK, CMV or EBV infection
* Recurrent pyelonephritis or need for indwelling or self-catheterization
* Prior amputation or ischemic rest pain
* Women who are pregnant, nursing, or who plan to become pregnant whilst in the trial.
* History of pancreatitis
* Personal or family history or medullary thyroid cancer or MEN2B
* History of unstable diabetic retinopathy within 1 year prior to screening
* Use of SGLT2i or GLP-1RA within 30 days prior to screening.
* Current and frequent episodes of hypoglycemia
* Current history of DKA requiring medical intervention or hospitalization
* With current risk of volume depletion, hypotension and/or electrolyte imbalance
* With known or suspected hypersensitivity to semaglutide or related products
* Patient not able to understand and comply with study requirements, based on Investigator's judgment.
* Any other clinical condition that, based on Investigator's judgement, would jeopardize patient safety during trial participation or would affect the study outcome (e.g. immunocompromised patients, active malignancy, patients who might be at higher risk of developing genital or mycotic infections, patients with chronic viral infections, uncontrolled hypertension, cardiorenal and/or hepatorenal syndrome etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Proximal tubular natriuresis with combination therapy | From baseline to combination therapy end (24 weeks)
  Measured by fractional excretion of sodium
Proximal tubular natriuresis with monotherapy | From baseline to monotherapy end (12 weeks)
  Measured by fractional excretion of sodium

SECONDARY OUTCOMES:
Measured Glomerular Filtration Rate | From baseline to monotherapy end (12 weeks) and combination therapy end (24 weeks) ]
  GFR, based on plasma iohexol clearance
Estimated Glomerular Filtration Rate | From baseline to monotherapy end (12 weeks) and combination therapy end (24 weeks) ]
  GFR, based on serum creatinine
Urinary 8-hydroxydeoxyguanosine and 8-isoprostane concentration | From baseline to monotherapy end (12 weeks) and combination therapy end (24 weeks) ]
  Using ELISA
Urinary albumin excretion | From baseline to monotherapy end (12 weeks) and combination therapy end (24 weeks) ]
  From 24-hour urine collection
Arterial stiffness | From baseline to monotherapy end (12 weeks) and combination therapy end (24 weeks) ]
  Measured using a Sphygmocor device
Liver stiffness | From baseline to monotherapy end (12 weeks) and combination therapy end (24 weeks) ]
  Using transient elastography
Diastolic function | From baseline to monotherapy end (12 weeks) and combination therapy end (24 weeks) ]
  Using 2D echocardiography
Change in percentage of glycated hemoglobin (HbA1c) | From baseline to monotherapy end (12 weeks) and combination therapy end (24 weeks) ]
Change in concentration of urine glucose excretion | From baseline to monotherapy end (12 weeks) and combination therapy end (24 weeks) ]
  Urinary analysis will be performed to quantify the amount of glucose excretion.
Change in body composition (percent body mass, body fat, and muscle mass) | From baseline to monotherapy end (12 weeks) and combination therapy end (24 weeks) ]
  Bioimpedence measurements will be taken to study the effects of intervention on body composition.
Change in body weight | From baseline to monotherapy end (12 weeks) and combination therapy end (24 weeks) ]
Safety: the incidence of acute kidney injury. | From baseline to monotherapy end (12 weeks) and combination therapy end (24 weeks) ]
Safety: the incidence of hypotension | From baseline to monotherapy end (12 weeks) and combination therapy end (24 weeks) ]
Safety: The incidence of hyperkalemia | From baseline to monotherapy end (12 weeks) and combination therapy end (24 weeks) ]
Safety: The incidence of urinary and mycotic infections. | From baseline to monotherapy end (12 weeks) and combination therapy end (24 weeks) ]
Safety: The number of ketoacidosis events. | From baseline to monotherapy end (12 weeks) and combination therapy end (24 weeks) ]
Safety: The incidence of amputations. | From baseline to monotherapy end (12 weeks) and combination therapy end (24 weeks) ]
Safety: The incidence of pancreatitis or biliary complications | From baseline to monotherapy end (12 weeks) and combination therapy end (24 weeks) ]
Safety: The number of allergic reaction events. | From baseline to monotherapy end (12 weeks) and combination therapy end (24 weeks) ]

CONTACTS AND LOCATIONS:
Overall Officials: Sunita Singh, MD MSc FRCPC, Principal Investigator — University Health Network, Toronto General Hospital
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No